CLINICAL TRIAL: NCT03636009
Title: The Concurrent Use of Intermittent Cervical Traction and Neuromobilization Techniques in Patients With Cervical Radiculopathy
Brief Title: Concurrent Treatment for Patients With Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Indianapolis (Other)
Responsible Party: Principal Investigator, James W. Bellew, Professor, University of Indianapolis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0924
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Spinal Nerve Root Disorder Nos
Keywords: cervical radiculopathy; neck pain; neuromobilizations
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Intervention Model Description: Two groups receiving interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent traction (Experimental): Concurrent traction and neuromobilization technique at each scheduled session Active exercise program (4-5 exercises) at each session Manual therapy to cervical and thoracic spine at each session
  Interventions: Other: concurrent traction and neuromobilization technique; Other: active exercise program; Other: manual therapy to cervical and thoracic spine
- Sequential traction (Active Comparator): Sequential traction and neuromobilization technique at each scheduled session Active exercise program (4-5 exercises) at each session Manual therapy to cervical and thoracic spine at each session
  Interventions: Other: sequential traction and neuromobilization technique; Other: active exercise program; Other: manual therapy to cervical and thoracic spine

INTERVENTIONS:
Other: concurrent traction and neuromobilization technique — participant will be on a mechanical traction machine with an on:off cycle. During the on cycle, the primary researcher will be performing a neuromobilization technique on the symptomatic arm. Patients will also receive exercise and manual therapy
  Other Names: Concurrent traction; Neurmobilization technique
  Arms: Concurrent traction
Other: sequential traction and neuromobilization technique — Participants will receive neuromobilzation techniques followed by supine cervical traction
  Other Names: Sequential traction
  Arms: Sequential traction
Other: active exercise program — Participants will have 4-5 exercises to perform at each session
Other: manual therapy to cervical and thoracic spine — Lateral glides to cervical spine and thoracic manipulations

SUMMARY:
This study evaluates the effectiveness of two treatment interventions in patients with cervical radiculopathy. One group will receive a concurrent approach using traction and neuromobilizations. The other group will receive the sequential approach of traction and neuromobilizations

DETAILED DESCRIPTION:
Physical therapists routinely use cervical traction and manual therapy in patients with cervical radiculopathy. The standard of care is a sequential approach in which the patients receive interventions successively. This study will provide the standard of care approach for one group while the other group receives the concurrent approach in which the patient will have neuromobilizations while they are receiving mechanical traction. Both groups will also receive exercise and manual therapy to the cervical and thoracic spine.

ELIGIBILITY:
Inclusion criteria:

* Participants that test positive on at least 3 out of 4 special tests.
* Participants will score at least 10 on the Neck Disability Index
* Participants will score at least 2 on the numeric pain rating scale

Exclusion Criteria:

* Do not test positive on at least 3 of 4 special tests.
* Signs of cervical trauma
* Cervical myelopathy
* Active pregnancy
* Medical red flags (fracture, tumor, long term steroid use, rheumatoid arthritis, and osteoporosis)
* Evidence of vascular compromise
* Cervical spine surgery
* Recent injections in the past six weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
changes in pain | after 4 weeks of intervention
  Measured using the Numeric pain rating scale. Minimum score is 0 and maximum score is 10. 0 describes no pain and 10 describes worst pain imaginable.
changes in function | After 4 weeks of intervention
  Measured using the Neck Disability Index. The Neck Disability Index has a minimum score of 0 and maximum score of 50. It is typically expressed as a percentage by multiplying the score by 2. Higher scores represent greater disability.

SECONDARY OUTCOMES:
Difference in treatment time between the groups | 4 weeks of intervention
  average minutes in treatment in each group

CONTACTS AND LOCATIONS:
Overall Officials: James Bellew, EdD, Principal Investigator — University of Indianapolis
Locations (1):
- Michiana Orthopaedics and Sports Physical Therapy, Mishawaka, Indiana, United States

IPD SHARING:
Plan to Share IPD: No